CLINICAL TRIAL: NCT04912908
Title: Validation of a Surgical Navigation Algorithm During Knee Replacements in Patients With Knee Osteoarthritis
Acronym: VALALGON
Status: Completed | Type: Observational
Sponsor: Ganymed Robotics (Industry)
Responsible Party: Sponsor
Other Study IDs: 2021-A00961-40
Record Dates: First submitted 2021-06-02; First posted 2021-06-03 (Actual); Last update posted 2022-11-18 (Actual); Status verified 2022-11

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Images taken during knee replacement surgery — Images taken during knee replacement surgery will be compared to CT-Scan that was performed before surgery
  Other Names: CT-Scan before knee replacement surgery

SUMMARY:
Ganymed Robotics develops a novel solution of surgical navigation to assist surgeons during knee remplacement surgeries. The aim of this study is to train and validate this novel algorithm.

DETAILED DESCRIPTION:
During knee replacement surgery, per-operative images of the patient's knee will be taken. These images will then be compared with the pre-operative CT-scan of the patient using the novel navigation algorithm. The algorithm will be validated based on its ability to correctly compare both modalities (pre-operative and per-operative images).

ELIGIBILITY:
Inclusion Criteria:

* Adults patients who signed the ICF of the study
* Patients suffering from knee osteoarthritis requiring a total knee replacement surgery

Exclusion Criteria:

* Patient under the age 18
* Patient unable to consent to the study or refusing to participate
* Patient with history of knee replacement on the knee that will be operated again
* Patient unable to realize a pre-operative CT-scan
* Patient not covered by French Health insurance or equivalent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The surgeons involved in the study will propose to all patients corresponding to the eligibility criteria to participate to the study during pre-surgery appointment.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-07-07 (Actual); Primary Completion 2022-07-08 (Actual); Study Completion 2022-07-08 (Actual)

PRIMARY OUTCOMES:
Validation of navigation algorithm | 12 months
  Comparison between peroperative images and preoperative CT-scan

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital prive Jean Mermoz-Ramsay Santé, Lyon, France

IPD SHARING:
Plan to Share IPD: No